CLINICAL TRIAL: NCT03361865
Title: A Phase 3 Randomized, Double-Blind Trial of Pembrolizumab (MK-3475) in Combination With Epacadostat (INCB024360) or Placebo in Participants With Cisplatin-ineligible Urothelial Carcinoma (KEYNOTE-672/ECHO-307)
Brief Title: Pembrolizumab in Combination With Epacadostat or Placebo in Cisplatin-ineligible Urothelial Carcinoma (KEYNOTE-672/ECHO-307)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEYNOTE-672/ECHO-307; 2017-002311-34 (EudraCT Number)
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Results first posted 2019-08-29 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: UC (Urothelial Cancer)
Keywords: Urothelial cancer, programmed cell death 1 (PD-1) inhibitor; indoleamine 2,3-dioxygenase (IDO) inhibitor
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Masking Description: The study will be unblinded after the last participant completes Week 9 imaging assessment for efficacy analysis and after appropriate EC/IRB approvals have been received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab 200 mg + epacadostat 100 mg BID (Experimental): Pembrolizumab + epacadostat
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat
- Pembrolizumab 200 mg + placebo BID (Active Comparator): Pembrolizumab + placebo
  Interventions: Drug: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administered intravenously every 3 weeks.
  Other Names: MK-3475
Drug: Epacadostat — Epacadostat administered orally twice daily.
  Other Names: INCB024360
  Arms: Pembrolizumab 200 mg + epacadostat 100 mg BID
Drug: Placebo — Matching placebo administered orally twice daily.
  Arms: Pembrolizumab 200 mg + placebo BID

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of pembrolizumab + epacadostat vs pembrolizumab + placebo in participants with cisplatin-ineligible urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed diagnosis of advanced/unresectable (inoperable) or metastatic urothelial cancer of the renal pelvis, ureter, bladder, or urethra.
* Measurable disease based on RECIST v1.1.
* Be considered ineligible to receive cisplatin-based combination therapy, based on protocol-defined criteria.
* Have provided tissue for PD-L1 analysis from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
* Have received no prior systemic chemotherapy for advanced/unresectable (inoperable) or metastatic urothelial cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 within 14 days prior to randomization.
* Adequate organ function per protocol-defined criteria.

Exclusion Criteria:

* Disease that is suitable for local therapy administered with curative intent.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, ie, without evidence of progression for at least 4 weeks by repeat imaging, clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* Known history of human immunodeficiency virus (HIV) infection. HIV testing is not required unless mandated by local health authority.
* Known history of or is positive for active hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or has active hepatitis C (HCV RNA). Note: Testing must be performed to determine eligibility.
* History of a gastrointestinal condition that in the opinion of the Investigator may affect oral drug absorption.
* History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful.
* Use of protocol-defined prior/concomitant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2020-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jones, MD, Study Director — Incyte Corporation
Locations (143):
- United States (22):
  - Arizona Oncology Associates PC- HOPE, Tucson, Arizona
  - University of California Irvine Medical Center, Orange, California
  - Yale Cancer Center, New Haven, Connecticut
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - GU Research Network-Urology Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina-Hollings Cancer Center, Charleston, South Carolina
  - Tennessee Oncology, PLLC/The Sarah Cannon Research Institute, Chattanooga, Tennessee
  - University of Tennessee Medical Center Knoxville, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology-Memorial City, Houston, Texas
  - University of Washington, Seattle, Washington
- Australia (5):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Austin Health-Austin Hospital, Heidelberg, Victoria
  - Adelaide Cancer Centre, Kurralta Park
  - Macquarie University Hospital, Macquarie Park
- Belgium (7):
  - Institut Jules Bordet, Brussels
  - Grand Hopital de Charleroi - Site Notre Dame - Oncology, Charleroi
  - AZ Maria Middelares Gent, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - AZ Nikolaas, Sint-Niklaas
  - GZA Sint Augustinus, Wilrijk
- Canada (6):
  - Moncton Hospital - Horizon Health Network, Moncton, New Brunswick
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHU de Quebec - Hotel-Dieu de Quebec, Québec, Quebec
- France (13):
  - Institut de Cancerologie de l Ouest Site Paul Papin, Angers
  - CHU de Besancon, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Paoli Calmettes, Marseille
  - Centre d Oncologie de Gentilly, Nancy
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - CHU de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - C.H.U. de Tours - Hopital Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Universitaetsklinikum Schleswig-Holstein. Campus Luebeck, Lübeck, Schleswig-Holstein
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Kliniken Essen Mitte, Essen
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Magdeburg A.o.R., Magdeburg
  - Klinikum rechts der Isar der Technischen Universitat, München
  - Krankenhaus der Barmherzigen Brueder Trier, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
- Ireland (5):
  - Cork University Hospital, Cork
  - Adelaide & Meath Hospital (Incl NCH), Dublin
  - University College Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford
- Israel (7):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (6):
  - Medical Oncology Ospedale San Donato, Arezzo
  - Istituto Tumori Giovanni Paolo II, Bari
  - Istituto Scientifico Romagnolo per Studio e Cura Tumori IRST, Meldola
  - Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto, Padua
- Japan (9):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Nara Medical University Hospital, Kashihara, Nara
  - Kindai University Hospital, Sayama, Osaka
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Tokushima University Hospital, Tokushima
  - Medical Hospital, Tokyo Medical And Dental University, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Netherlands (6):
  - Amphia Ziekenhuis, Breda, North Brabant
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - VU University Medical Center, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - University Medical Center Groningen, Groningen
  - Erasmus MC, Rotterdam
- Poland (9):
  - Beskidzkie Centrum Onkologii im. Jana Pawla II, Bielsko-Biala
  - Wojewodzkie Centrum Szpitalne Kotliny Jeleniogorskiej, Jelenia Góra
  - Uniwersyteckie Centrum Kliniczne Slaskiego Uniwersytetu Medycznego, Katowice
  - GLOBE Badania Kliniczne Oddzial we Wroclawiu, Komorowice
  - Europejskie Centrum Zdrowia Otwock, Otwock
  - Urologica Praktyka Lekarska Adam Marcheluk, Siedlce
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM w Szczecinie, Szczecin
  - Magodent Szpital Elblaska, Warsaw
  - Szpital Sw. Elzbiety Mokotowskie Centrum Medyczne, Warsaw
- Russia (8):
  - Leningrad Regional Oncology Dispensary, Saint Petersburg, Leningrad Region, Vsevolozhsky District
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - N.N. Blokhin NMRCO, Moscow
  - Russian Scientific Center of Roentgenoradiology, Moscow
  - National Medical Research Radiological Centre, Moscow
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - Pokrovskaya City Hospital, Saint Petersburg
  - Clinic of Bashkortostan State Medical University, Ufa
- South Korea (5):
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital Teresa Herrera - Chuac, A Coruña
  - Hospital Infanta Cristina, Badajoz
  - Hospital General Universitari Vall d Hebron, Barcelona
  - ICO L Hospitalet, L'Hospitalet de Llobregat
  - Hospital Universitario Lucus Augusti, Lugo
  - Xarxa Assistencial Universitaria Manresa, Manresa
  - Consorci Hospitalari Parc Tauli de Sabadell, Sabadell
  - Hospital Virgen del Rocio, Seville
- Taiwan (5):
  - Taipei Veterans General Hospital, Taipei, Beitou
  - Chang Gung Medical Foundation - Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Ukraine (6):
  - MI Dnipr Regional Clinical Hospital named after I.I. Mechnikov, Dnipropetrovsk
  - Dnipropetrovsk City Multidiscipline Clinical Hosp.4 of DRC, Dnipropetrovsk
  - Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Kyiv City Clinical Oncology Center, Kyiv
  - MI Odessa Regional Oncological Centre, Odesa
  - RMI Sumy Regional Clinical Oncology Dispensary, Sumy
- United Kingdom (7):
  - Royal Marsden NHS Trust, Sutton, Surrey
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Barts Health NHS Trust - St Bartholomew's Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Plymouth Hospitals NHS Trust, Plymouth
  - Sunderland Royal Hospital, Sunderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Necchi A, Van der Heijden MS, Trukhin D, Peer A, Gurney H, Alekseev BY, Parnis FX, Leibowitz R, De Santis M, Grivas P, Clark J, Munteanu M, Kataria R, Jia C, Balar AV, de Wit R. Pembrolizumab plus either epacadostat or placebo for cisplatin-ineligible urothelial carcinoma: results from the ECHO-307/KEYNOTE-672 study. BMC Cancer. 2024 Jul 25;23(Suppl 1):1252. doi: 10.1186/s12885-023-10727-3. PMID 39054491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 47 centers in 15 countries.
Groups:
- Pembrolizumab 200 mg + Epacadostat 100 mg BID: Pembrolizumab administered intravenously every 3 weeks. Epacadostat administered orally twice daily.
- Pembrolizumab 200 mg + Placebo BID: Pembrolizumab administered intravenously every 3 weeks. Matching placebo administered orally twice daily.
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID
Started | 44 | 49
Intention-to-Treat (ITT) | 44 | 49
All Participants as Treated (APaT) | 43 | 49
Completed (Refers to participants that discontinued study with amendment 4, and didn't require follow-up.) | 25 | 22
Not Completed | 19 | 27
Not completed — Death | 17 | 18
Not completed — Physician Decision | 1 | 9
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID | Total
Number analyzed (Participants) | 44 | 49 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (9.5) | 72.4 (8.9) | 72.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 33 | 38 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 35 | 42 | 77
  Unknown or Not Reported | 7 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9 | 8 | 17
  White | 33 | 37 | 70
  Missing | 2 | 4 | 6
Metastasis Status at Screening [Count of Participants; unit: Participants]
  Metastatic | 38 | 45 | 83
  Advanced/Unresectable | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) With Pembrolizumab + Epacadostat Versus Pembrolizumab + Placebo
Description: ORR was defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR) per RECIST v1.1 by investigator determination. Responses are based on Investigator assessments per RECIST 1.1 without confirmation using all scans up to the cutoff date.
Time Frame: Week 9
Population: The Intention-to-Treat (ITT) population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID
Number analyzed (Participants) | 44 | 49
percentage of participants | 31.8 [22.46 to 55.24] | 24.5 [15.33 to 43.67]

2. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Epacadostat Versus Pembrolizumab + Placebo as Measured by Number of Participants Experiencing Adverse Events (AEs)
Description: AE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to approximately 25 months
Population: All Participants as Treated (APaT) population consisted of all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID
Number analyzed (Participants) | 43 | 49
Participants | 43 | 47

3. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Epacadostat Versus Pembrolizumab + Placebo as Measured by Number of Participants Discontinuing Study Treatment Due to AE
Description: as for outcome 2
Time Frame: Up to approximately 25 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID
Number analyzed (Participants) | 43 | 49
Participants | 11 | 15

ADVERSE EVENTS:
Time Frame: up to approximately 25 months
Description: The All Participants as Treated (APaT) population was used for the safety analysis and consisted of all randomized participants who received at least 1 dose of study treatment. All-Cause Mortality was based on the ITT population and consisted of all randomized participants. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the drug are excluded.
Groups:
- Total: Total
Arm/Group | Pembrolizumab 200 mg + Epacadostat 100 mg BID | Pembrolizumab 200 mg + Placebo BID | Total
All-Cause Mortality (participants affected / at risk) | 17/43 | 19/49 | 36/92
Serious Adverse Events (participants affected / at risk) | 23/43 | 23/49 | 46/92
Other Adverse Events (participants affected / at risk) | 42/43 | 47/49 | 89/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg + Epacadostat 100 mg BID (N=43) | Pembrolizumab 200 mg + Placebo BID (N=49) | Total (N=92)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 3 (4) | 3 (4)
Death (General disorders) | 1 (1) | 1 (1) | 2 (2)
Device occlusion (Product Issues) | 2 (2) | 0 (0) | 2 (2)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Huntington's disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 5 (5) | 13 (14)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 6 (10) | 9 (13)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 1 (2) | 3 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg + Epacadostat 100 mg BID (N=43) | Pembrolizumab 200 mg + Placebo BID (N=49) | Total (N=92)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (6) | 8 (8)
Alanine aminotransferase increased (Investigations) | 4 (4) | 5 (7) | 9 (11)
Amylase increased (Investigations) | 4 (8) | 4 (4) | 8 (12)
Anaemia (Blood and lymphatic system disorders) | 14 (14) | 9 (12) | 23 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (5) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 5 (6) | 9 (10)
Asthenia (General disorders) | 9 (9) | 10 (10) | 19 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (9) | 15 (16)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 5 (5) | 7 (7)
Blood creatinine increased (Investigations) | 5 (6) | 3 (6) | 8 (12)
Constipation (Gastrointestinal disorders) | 7 (10) | 7 (7) | 14 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6) | 9 (10)
Creatinine renal clearance decreased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 5 (7) | 8 (8) | 13 (15)
Diarrhoea (Gastrointestinal disorders) | 10 (14) | 7 (9) | 17 (23)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 8 (8)
Dysuria (Renal and urinary disorders) | 3 (3) | 3 (3) | 6 (6)
Fatigue (General disorders) | 6 (7) | 8 (9) | 14 (16)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 4 (4)
Haematuria (Renal and urinary disorders) | 4 (5) | 7 (9) | 11 (14)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (6) | 7 (9)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (7) | 0 (0) | 3 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 7 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 3 (4)
Hypothyroidism (Endocrine disorders) | 3 (3) | 4 (4) | 7 (7)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 5 (5)
Lipase increased (Investigations) | 4 (4) | 4 (4) | 8 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (9) | 6 (6) | 12 (15)
Oedema peripheral (General disorders) | 3 (4) | 7 (10) | 10 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 5 (5)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (13) | 6 (7) | 16 (20)
Pyrexia (General disorders) | 5 (6) | 6 (8) | 11 (14)
Rash (Skin and subcutaneous tissue disorders) | 10 (12) | 14 (14) | 24 (26)
Urinary tract infection (Infections and infestations) | 5 (5) | 11 (14) | 16 (19)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (9) | 11 (13)
Weight decreased (Investigations) | 3 (3) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT03361865/Prot_SAP_000.pdf